CLINICAL TRIAL: NCT04279873
Title: Use of Microscopy, Cultures and Molecular Biological Methods for Diagnosing Nosocomial Pneumonia in Patients Admitted to the Intensive Care Unit - an Exploratory Study
Brief Title: Use of Microscopy, Cultures and Molecular Biological Methods for Diagnosing Nosocomial Pneumonia
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Collaborators: Slagelse Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REG-048-2014; REG-48-2017 (Other: The Danish Data Protection Agency)
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Nosocomial Pneumonia
Keywords: Nosocomial, Pneumonia; Diagnostics; 16s; 18s; PCR; Next Generation Sequencing
MeSH Terms: conditions — Healthcare-Associated Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pulmonary secretion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with nosocomial pneumonia: Diagnostic procedures on pulmonary secretion collected by tracheal suctioning and bronchoalveolar lavage.
  Interventions: Diagnostic Test: Microbiological diagnostics on pulmonary secretion

INTERVENTIONS:
Diagnostic Test: Microbiological diagnostics on pulmonary secretion — Culture, 16s, 18s, next generation sequencing

SUMMARY:
Nosocomial pneumonia in the Intensive Care Unit is often not properly diagnosed mainly due to ongoing antimicrobial therapy. The study investigates the feasibility of more advanced diagnostic technics.

DETAILED DESCRIPTION:
ICU patients fulfilling the CDC criteria for nosocomial pneumonia and mechanically ventilated for no more than 24 hours are included in the study. The material for the diagnostic procedure is pulmonal secretion collected by 1. suctioning in the tracheal tube and 2. bronchioalveolar lavage. The diagnostic procedures are culturing, 16S and18S gene PCR and subsequent sequencing. The 3 diagnostic methods will be compared in order of proper diagnosis and the ability to determine a specific antimicrobial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients intubated because of respiratory failure following nosocomial pneumonia

Exclusion Criteria:

* Terminal patients
* Patients with lung cancer
* Intubated for more than 24 hours at the sampling time
* Not fulfilling the CDC criteria for nosocomial pneumonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with nosocomial pneumonia and the need of mechanical ventilation not intubated for more than 24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Ratio of patients where the advanced methods are superior to routine | 1 day
  Ratio of patients diagnosed by 16s, 18s or NGS to total number of patients compared to ratio of patients diagnosed by routine method (culture)

CONTACTS AND LOCATIONS:
Overall Officials: Lone Musaeus Poulsen, MD, Principal Investigator — Zealand University Hospital
Locations (1):
- Zealand University Hospital, Køge, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No